CLINICAL TRIAL: NCT06023784
Title: The Impact of Left Bundle Branch Area Pacing Versus Right Ventricular Pacing on the Incidence of New-onset Atrial Fibrillation in Patients With Atrioventricular Block: a Randomized Controlled Trial
Brief Title: The Impact of LBBAP vs RVP on the Incidence of New-onset Atrial Fibrillation in Patients With Atrioventricular Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: the July study
Record Dates: First submitted 2023-08-24; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-07

CONDITIONS: Left Bundle Branch Area Pacing; Right Ventricular Pacing; Atrioventricular Block; Atrial Fibrillation
MeSH Terms: conditions — Atrioventricular Block; Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left bundle branch area pacing (Experimental)
  Interventions: Procedure: left bundle branch area pacing
- right ventricular pacing (Active Comparator)
  Interventions: Procedure: right ventricular pacing

INTERVENTIONS:
Procedure: left bundle branch area pacing — Left bundle branch area pacing(LBBAP) is a novel physiological pacing form for ventricular pacing. In patients received LBBAP, the pacing lead will be placed at left bundle branch area to achieve narrow paced QRS duration.
  Arms: left bundle branch area pacing
Procedure: right ventricular pacing — Right ventricular pacing is the traditional pacing modality for ventricular pacing. The pacing lead was placed in the apex or septum of right ventricle.
  Arms: right ventricular pacing

SUMMARY:
This is a single-center, randomized controlled study. The aim of this study is to compare the impact of left bundle branch area pacing versus traditional right ventricular pacing on the incidence of atrial fibrillation in patients with atrioventricular block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-85;
* AV block patients with ventricular pacing indications and the expected rate of ventricular pacing(VP)> 40%, including (a) third-degree AV block; (b) second degree AV block (type II); (c) intermittent advanced AV block with expected VP>40%; (d) symptomatic first degree AV block and PR interval on ECG > 300ms;
* Signed informed consent;

Exclusion Criteria:

* Baseline echocardiographic assessment of patients with impaired LV function (LVEF<50%);
* Patients with the history of atrial fibrillation;
* Having difficulties in follow-up: Those who cannot accept 2-year follow-up on time due to physical condition or other reasons;
* Pacemaker replacement without new implanted ventricular electrodes;
* Surgery is required within 1 year due to severe structural heart disease;
* Patients with tricuspid mechanical valve replacement, or congenital heart disease (including transposition of the great arteries, or permanent left superior vena cava, etc);
* AV block resulting from: (a) Hypertrophic cardiomyopathy(HCM), (b) ventricular septal defect repair, and those who are unlikely to achieve successful LBBAP procedure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of new-onset atrial fibrillation | within two years after device implantation

SECONDARY OUTCOMES:
all-cause mortality | within two years after device implantation
hospitalization for heart failure | within two years after device implantation
an device upgrade for heart failure | within two years after device implantation
alteration of quality of life score | within two years after device implantation
Improvement of left ventricular, right ventricular and left atrial function measured by echocardiography | within two years after device implantation
pacemaker-associated cardiomyopathy | within two years after device implantation

CONTACTS AND LOCATIONS:
Overall Officials: Taibo Chen, PhD., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No